CLINICAL TRIAL: NCT04190017
Title: Comparison of Brain Volumes of Preterm Infants Measured by Two Dimensional Ultrasonography and Cranial Magnetic Resonance Imaging
Brief Title: Comparison of Brain Volumes Measured by 2D USG and MRI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Fuat Emre Canpolat, Assoc Prof Fuat Emre CANPOLAT MD, Ankara City Hospital Bilkent
Other Study IDs: 2019512-1
Record Dates: First submitted 2019-12-05; First posted 2019-12-09 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Central Nervous System Vulnerabilities in Preterm Infants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Cranial MRI — Cranial MRI

SUMMARY:
Cranial USG is simple and easy method to assess preterm infant brain. Some studies showed that brain volumes of preterm infants could be calculated by measurement of 2D distances. Our aim in this study was to compare brain volume obtained by USG and MRI.

DETAILED DESCRIPTION:
All preterm infants less than 32 weeks of gestational age undergo cranial USG examination routinely at least, in the first week of life, at the end of first month and corrected age 36 weeks and 40 weeks. We will performa all USG mesurements with measureing intracranial hegiht, anteroposterior diameter, biparietal diamater, ventriccular height, thalamo-occipital distance and ventricular index. We will calculate the brain volume as a spheric geometric shape than we will calculate two ventricles as conical shapes. Absolute brain volume will be calculating by substracting two ventricles from total brain volume. At 40 weeks of age we will perform a cranial MRI to show exact brain volume and we will ccompare two different methods.

ELIGIBILITY:
Inclusion Criteria:

* All preterm infants under 32 weeks of gestational age and birth weight between 800-1200 grams
* Born in our hospital
* Alive during discharge

Exclusion Criteria:

* congenital anomalies
* cranial bleeding
* early death

Ages: 1 Day to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants under 32 weeks of GA and 800-1200 gram BW all admitted to Ankara Şehir Hospital MH5 NICU
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
Results of two different brain volumes | 6 months
  Patients in cohort will have both USG and cranial MRI

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Şenol Akın, MD, Study Chair — Ankara City Hospital Bilkent
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benavente-Fernandez I, Lubian-Gutierrez M, Jimenez-Gomez G, Lechuga-Sancho AM, Lubian-Lopez SP; Neonatal Neurology Foundation (Fundacion Nene). Ultrasound lineal measurements predict ventricular volume in posthaemorrhagic ventricular dilatation in preterm infants. Acta Paediatr. 2017 Feb;106(2):211-217. doi: 10.1111/apa.13645. Epub 2016 Nov 21. PMID 27783429
- [Background] Cheong JL, Thompson DK, Spittle AJ, Potter CR, Walsh JM, Burnett AC, Lee KJ, Chen J, Beare R, Matthews LG, Hunt RW, Anderson PJ, Doyle LW. Brain Volumes at Term-Equivalent Age Are Associated with 2-Year Neurodevelopment in Moderate and Late Preterm Children. J Pediatr. 2016 Jul;174:91-97.e1. doi: 10.1016/j.jpeds.2016.04.002. Epub 2016 May 9. PMID 27174146